CLINICAL TRIAL: NCT00018044
Title: Natural History, Genetics, Phenotype, and Treatment of Mycobacterial Infections
Brief Title: Study of Mycobacterial Infections
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Children's National Research Institute (Other); University of Miami (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010202; 01-I-0202
Record Dates: First submitted 2001-06-28; First posted 2001-06-29 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01-16

CONDITIONS: Mycobacterium Infections
Keywords: Mycobacterium Abscessus; Pulmonary; Mycobacterium Chelonae; Mycobacterium Avium Complex (MAC); Nontuberculous Mycobacteria (NTM); Natural History
MeSH Terms: conditions — Mycobacterium Infections; Mycobacterium Infections, Nontuberculous; Mycobacterium avium-intracellulare Infection | interventions — Clofazimine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Relatives: Blood relatives of enrolled patients
- Patients: Patients with mycobacterial infections
  Interventions: Drug: Clofazimine

INTERVENTIONS:
Drug: Clofazimine
  Groups: Patients

SUMMARY:
This study will examine the symptoms, course of disease and treatment of non-tuberculous mycobacterial (NTM) infections, as well as the genetics involved in these infections. Patients with NTM have recurrent lung infections and sometimes infections of the skin and other organs as well. They may also have curvature of the spine, barrel chest, and heart valve weakness. The study will compare the features of NTM with those of Job syndrome and cystic fibrosis, other diseases involving recurrent infections of the lungs and possibly other organs.

Patients with diagnosed or suspected non-tuberculous mycobacterial infection, cystic fibrosis or Job syndrome may be eligible for this study. All participants will have a medical and family history, blood and urine tests, imaging studies that may include X-rays, computed tomography (CT) or magnetic resonance imaging (MRI) scans, and DNA and other genetic studies. In addition, all patients with Job syndrome and cystic fibrosis, and patients with NTM who have lung disease undergo the following procedures:

* Scoliosis survey X-rays of the spine to look for curvature or other abnormalities of the spinal column
* Echocardiography imaging test that uses sound waves to examine the heart chambers and valves
* Electrocardiogram measurement of the electrical activity of the heart
* Pulmonary function tests breathing tests to measure how much air the patient can move into and out of the lungs
* Body measurements measurements of height, weight, arm span, finger length, etc.
* Joint function assessment of joint mobility using different maneuvers to test flexibility of joints and ligaments
* Examination of physical features that might be associated with NTM, such as high arched palate of the mouth, flat feet, or certain skin features
* Dermatology (skin) examination for reactive skin conditions or other skin problems and possibly a skin biopsy (surgical removal of a small skin tissue sample for microscopic examination)
* Interview with genetics specialist

These tests may require several days to complete. Patients with NTM will also be examined by a cystic fibrosis specialist and may have a sweat test. In addition, NTM patients will be asked to return to NIH every year for 5 years for follow-up tests, if medically indicated, including CT of the chest, scoliosis survey and examination by other specialists.

DETAILED DESCRIPTION:
The nontuberculous mycobacteria (NTM) are ubiquitous environmental organisms found in soil and water that rarely cause disease in humans. Since exposure to these organisms is universal and disease is rare, it can be concluded that normal host defenses are almost always sufficient to prevent infection. It follows that otherwise healthy individuals who develop disease must have abnormal susceptibility or immune defects that permit infection with nontubercuolous mycobacteria. The organisms that are most commonly encountered in clinical practice include Mycobacterium avium, and M. intracellulare [collectively known as the M. avium complex (MAC)], M. kansasii, M. fortuitum, M. abscessus, and M. chelonae. These organisms share significant structural and biochemical similarities with their more pathogenic relative, M. tuberculosis (MTB). Recognition of host factors that predispose or lead to NTM infection may have important implications for pathogenesis and therapeutic intervention, and may be applicable to the more virulent MTB. Identification of genetic or acquired susceptibility factors may lead to recognition of endogenous pathways that can be exploited therapeutically and to possible gene identification.

Over the last two decades, three important observations have been made regarding the pathogenesis of nontuberculous mycobacterial infections. 1) In patients infected with HIV, nontuberculous mycobacterial infections often occur when the CD4+ T-lymphocyte number falls below 50/mm3. This suggested that specific T cell products or activities were required for mycobacterial resistance. 2) An association was noted between pulmonary nontuberculous mycobacterial infections and a particular body habitus, predominantly in post-menopausal women (pectus excavatum, scoliosis, mitral valve prolapse). 3) Multiple defects have been found involving the interferon gamma synthesis and use pathways in patients with disseminated nontuberculous mycobacterial infection without HIV, suggesting this is a critical pathway for host defense against these organisms.

We seek to better characterize the predisposition to mycobacterial infection. This study will specifically address several aspects of immune function and investigate the proposed link to body morphotype in the relevant population. By collecting this information, we hope to provide insight into disease associations, infection susceptibility, and genetic predisposition to mycobacterial infection.

ELIGIBILITY:
* INCLUSION CRITERIA FOR PATIENTS:

This protocol will study patients with mycobacterial infections, including those without previously identified predisposing disease processes as well as individuals with underlying malignancies.

Patients with nontuberculous mycobacterial infections will be of particular interest, as we are interested in isolating and characterizing the primary immune defect(s) responsible for this infection susceptibility.

Select patients with acquired immunodeficiencies or tuberculosis may also be studied if relevant host defects are suspected.

Patients must be referred to NIH with a diagnosis or suspicion of having mycobacterial infection.

Male and female patients will be accepted without limitations due to age.

Only patients with nontuberculous mycobacterial infections without HIV infection will be considered for long-term disease management.

INCLUSION CRITERIA FOR RELATIVES:

As part of this protocol, we may obtain medical records, blood work, urine, saliva or buccal swab from some blood relatives of patients on the study, with the hope of isolating and characterizing the primary immune defect(s) responsible for mycobacterial infection susceptibilityand if there are any genetic links seen within families. We hope to identify families with an apparent genetic susceptibility to respiratory diseases predominantly associated with P-NTM and perform whole genome sequencing within this group to identify genetic mutations accounting for this increased susceptibility. Male and female patients will be accepted without limitation due to age. These relatives will not receive treatment or have any other protocol procedures done unless they become a patient on the study.

EXCLUSION CRITERIA:

None.

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with mycobacterial infections, including those without previously identified predisposing disease processes as well as individuals with underlying malignancies. Patients with nontuberculous mycobacterial infections will be of particular interest but select patients with acquired immunodeficiencies or tuberculosis may also be studied if relevant host defects are suspected. We may obtain specimens from some blood relatives of enrolled patients.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2001-01-01 (Actual)

PRIMARY OUTCOMES:
Collect patients with nontuberculous mycobacterial infections in order to identify known and novel immune defects, characterize the natural history of these infections in the setting of the best possible standard therapy, and explore the connect... | ongoing
  Collecting information on mycobacterial infections

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Holland, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] West RR, Hsu AP, Holland SM, Cuellar-Rodriguez J, Hickstein DD. Acquired ASXL1 mutations are common in patients with inherited GATA2 mutations and correlate with myeloid transformation. Haematologica. 2014 Feb;99(2):276-81. doi: 10.3324/haematol.2013.090217. Epub 2013 Sep 27. PMID 24077845
- [Derived] Purisch SE, Shanis D, Zerbe C, Merideth M, Cuellar-Rodriguez J, Stratton P. Management of uterine bleeding during hematopoietic stem cell transplantation. Obstet Gynecol. 2013 Feb;121(2 Pt 2 Suppl 1):424-7. doi: 10.1097/aog.0b013e318270ecd3. PMID 23344397
- [Derived] Calvo KR, Vinh DC, Maric I, Wang W, Noel P, Stetler-Stevenson M, Arthur DC, Raffeld M, Dutra A, Pak E, Myung K, Hsu AP, Hickstein DD, Pittaluga S, Holland SM. Myelodysplasia in autosomal dominant and sporadic monocytopenia immunodeficiency syndrome: diagnostic features and clinical implications. Haematologica. 2011 Aug;96(8):1221-5. doi: 10.3324/haematol.2011.041152. Epub 2011 Apr 20. PMID 21508125
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2001-I-0202.html